CLINICAL TRIAL: NCT07241351
Title: Dexmedetomidine as an Adjunct to Fentanyl for Analgesia and Sedation of Term Neonates on Mechanical Ventilation
Brief Title: Dexmedetomidine as an Adjunct to Fentanyl for Term Neonates on Mechanical Ventilation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dexmedetomidine as an Adjunct
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Analgesia; Sedation and Analgesia; Neonatal; Mechanical Ventilation in Neonates
Keywords: sedation; analgesia; full term neonates; dexmedetomidine; fentanyl; adjuvant
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine and fentanyl (Experimental): fentanyl as a continuous infusion dose of 0.5 mcg/kg/hr over 24 hours with concomitant administration of DEX continuous IV infusion, over 24 hours, at a maintenance dose of 0.3 mcg/kg/hr for neonates <14 days and 0.5 mcg/kg/hr for those ≥14 days postnatal age
  Interventions: Drug: Dexmedetomidine; Drug: fentanyl 0.5 mcg/kg/hr
- fentanyl only (Active Comparator): fentanyl as continuous infusion at 1.0 mcg/kg/hr over 24
  Interventions: Drug: fentanyl 1mcg/kg/hr

INTERVENTIONS:
Drug: Dexmedetomidine — administration of DEX continuous IV infusion, over 24 hours, at a maintenance dose of 0.3 mcg/kg/hr for neonates <14 days and 0.5 mcg/kg/hr for those ≥14 days postnatal age
  Arms: dexmedetomidine and fentanyl
Drug: fentanyl 1mcg/kg/hr — fentanyl as continuous infusion at 1.0 mcg/kg/hr over 24 hours
  Arms: fentanyl only
Drug: fentanyl 0.5 mcg/kg/hr — fentanyl as a continuous infusion dose of 0.5 mcg/kg/hr over 24 hours with concomitant
  Arms: dexmedetomidine and fentanyl

SUMMARY:
Despite well conducted studies on pain management in mechanically ventilated neonates, there is still a need for exploration of appropriate and accurate pharmacological management strategies for this ongoing pain, and assessment of the clinical impact of the used drugs for analgesia and sedation.

In the current study, the aim was to reduce fentanyl doses on mechanical ventilated neonates after adding Dexmedetomidine

DETAILED DESCRIPTION:
Despite well conducted studies on pain management in mechanically ventilated neonates, there is still a need for exploration of appropriate and accurate pharmacological management strategies for this ongoing pain, and assessment of the clinical impact of the used drugs for analgesia and sedation. Opioids, such as fentanyl, are frequently used for analgesia and sedation in mechanically ventilated neonates with their short- and long-term adverse consequences Dexmedetomidine (DEX) is a specific alpha2 adrenergic agonist with promising data in NICU. Data exist that Dexmedetomidine recipient neonates require less adjunct sedation, experience less respiratory depression, less clinically significant hemodynamic effects, quicker establishment of enteral feeds and they could be extubated whilst on Dexmedetomidine infusion.

In the current study, the aim was to reduce fentanyl doses on mechanical ventilated neonates after adding Dexmedetomidine

ELIGIBILITY:
Inclusion Criteria:

* Full term neonates (≥ 37 weeks gestational age)
* Age: 1 to 28 days.
* Neonates just started invasive mechanical ventilation and are going to start sedation.

Exclusion Criteria:

* Presence of central nervous system abnormality
* Complex multiple congenital anomalies
* Neonates with facial malformations
* Neonates on mechanical Ventilation setting (peep above 9)

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
need for additional rescue analgesia | 24 hours
  number of doses of rescue analgesia given during the first 24 hours
NPASS ( neonatal pain , agitation and sedation score) | 24 hours
  done hourly to indicate pain and sedation if more than or equal to three patient is in pain

SECONDARY OUTCOMES:
development of bradycardia, | 24 hours
  development of bradycardia,
development of hypotension | 24 hours
  development of hypotension
development of respiratory depression | 24 hours
  development of respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: mariam JA ibrahim, PHD, Principal Investigator — Ain Shams University; Rouzan A Nassar, MBBCH, Principal Investigator — MOHP Egypt
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data can be shared from the corresponding author upon reasonable request
Supporting Information: Study Protocol